CLINICAL TRIAL: NCT02969252
Title: Pharmacokinetics and Safety Study of Rifamycin SV-MMX® 600 mg Tablets After Single and Multiple t.i.d. Doses in Healthy Male and Female Volunteers. Single and Multiple Dose, Open Label, Pharmacokinetics and Safety Study
Brief Title: Pharmacokinetics and Safety Study of Rifamycin SV-MMX® 600 mg Tablets After Single and Multiple t.i.d. Doses in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cosmo Technologies Ltd (Industry)
Responsible Party: Sponsor
Organization: CosmoTech (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CB-01-11/27
Record Dates: First submitted 2016-11-14; First posted 2016-11-21 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Healthy

ARMS (1):
- Open label (Other): Single and multiple dose, open label, pharmacokinetics and safety study
  Interventions: Drug: Rifamycin SV-MMX® 600

INTERVENTIONS:
Drug: Rifamycin SV-MMX® 600

SUMMARY:
The objective of the study was to evaluate the pharmacokinetics and the safety of rifamycin SV after single and multiple doses of Rifamycin SV-MMX® 600 mg tablets administered to male and female healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent: signed written informed consent before inclusion in the study
2. Sex and Age: men and women, 18-55 year old inclusive
3. Body Mass Index: 18.5-30 kgm2 inclusive
4. Vital signs: systolic blood pressure 100-139 mmHg, diastolic blood pressure 50-89 mmHg, heart rate 50-90 bpm, measured after 5 min at rest in the sitting position
5. Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the investigator and to comply with the requirements of the entire study
6. Fertility (women only): women of non-child-bearing potential or in post-menopausal status for at least 1 year.

For all female subjects, pregnancy test result had to be negative at screening and Day -1

Exclusion Criteria:

1. ECG 12-leads (supine position): clinically significant abnormalities
2. Physical findings: clinically significant abnormal physical findings which could interfere with the objectives of the study
3. Laboratory analyses: clinically significant abnormal laboratory values indicative of physical illness
4. Allergy: ascertained or presumptive hypersensitivity to the active principle and/or formulations' ingredients; history of anaphylaxis to drugs or allergic reactions in general, which the investigator considered could affect the outcome of the study
5. Diseases: significant history of renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, haematological, endocrine or neurological diseases that could interfere with the aim of the study
6. Medications: medications, including over the counter medications and herbal remedies, for 2 weeks before the start of the study
7. Investigative drug studies: participation in the evaluation of any investigational product for 3 months before this study. The 3-month interval was calculated as the time between the first calendar day of the month that follows the last visit of the previous study and the first day of the present study
8. Blood donation: blood donations for 3 months before this study
9. Drug, alcohol, caffeine, tobacco: history of drug, alcohol (more than 1 drink a day for females and more than 2 drinks a day for males, defined according to the USDA Dietary Guidelines 2010), caffeine (more than 5 cups coffee/tea/day) or tobacco abuse (10 cigarettes a day)
10. Abuse drug test: positive result at the drug test at screening or Day-1
11. Alcohol test: positive alcohol breath test at Day -1
12. Diet: abnormal diets (less than1600 or more than 3500 kcal/day) or substantial changes in eating habits in the 4 weeks before this study; vegetarians
13. Pregnancy (females only): positive or missing pregnancy test at screening or Day -1, pregnant or lactating women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-07; Primary Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Cmax | Day 1
  Cmax,0-24 h
Cmax | Day 1
  Cmax,0-6
tmax | Day 1
  tmax,0-24
tmax | Day 1
  tmax,0-6
AUC | Day 1
  AUC 0-24
AUC | Day 1
  AUC 0-6

REFERENCES:
- [Derived] Di Stefano AFD, Radicioni MM, Vaccani A, Mazzetti A, Longo LM, Moro L. Pharmacokinetics and Safety of Rifamycin SV after Single and Multiple Doses of MMX(R) Modified Release Tablets in Healthy Male and Female Volunteers. Antibiotics (Basel). 2021 Feb 6;10(2):167. doi: 10.3390/antibiotics10020167. PMID 33562091